CLINICAL TRIAL: NCT07199985
Title: Assessment of Intrinsic Risk Factors for Ankle Injuries in Ballet Dancers
Status: Active, not recruiting | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Erdem Engin, Resident at department of sports medicine, Ege University
Other Study IDs: 25-10T/15
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Ballet dancers; ankle injuries; isokinetic strength; intrinsic risk
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ballet dancers without ankle injury: Ankle muscle isokinetic strength, joint range of motion, and dynamic and static balance will be measured in ballet dancers who have not taken a break from dancing in the last 12 months.
- Ballet dancers with ankle injury: The isokinetic strength of the ankle muscles, joint range of motion, and dynamic and static balance of ballet dancers who have taken at least a week off from dancing due to an ankle injury within the last 12 months will be measured.
- Control: The ankle isokinetic muscle strength, joint range of motion, dynamic and static balance of healthy male and female volunteers over the age of 18 without ankle injuries will be measured.

SUMMARY:
This study aims to evaluate intrinsic risk factors (muscle strength, joint range of motion, static and dynamic balance) that may lead to ankle injuries in ballet dancers and to examine the relationship between these factors and ankle injuries experienced in the last 12 months. By comparing ballet dancers who have suffered injuries requiring physical therapy or forcing them to take a break from dancing for more than one week in the past year with uninjured ballet dancers and a control group, the findings aim to contribute scientifically to the development of individualized rehabilitation programs and the safe and effective planning of return-to-stage processes. Furthermore, it is believed that these data may support the reduction of time and financial losses among dancers.

DETAILED DESCRIPTION:
This study aims to evaluate intrinsic risk factors that may lead to ankle injuries in ballet dancers. Ankle injury risk factors are divided into two categories: intrinsic and extrinsic. Extrinsic risk factors are external to the individual, such as surface type, shoe wear, and type of athletic activity (training and competition) that may affect the athlete's performance. Intrinsic risk factors include age, gender, strength, joint range of motion, balance, and motor control, which affect the athlete's ability to perform sports-related activities. The study will be conducted with a total of 45 participants, including 30 participants aged 18 and over who reside in Izmir and are professional ballet dancers, and 15 control participants who have no previous dance experience. Of the 30 professional ballet dancers, 15 will be selected from dancers who have suffered an ankle injury requiring physical therapy or forcing them to take at least a one-week break from the stage within the last year. The other 15 ballet dancers will be those who have not experienced any problems due to an ankle injury within the last year. Participants will be asked whether they have suffered an injury requiring medical attention in the ankle region within the last 12 months; the data obtained will be correlated with various biomechanical measurements. Each participant will perform a standard warm-up program before the tests.

The four main parameters to be evaluated in the study are as follows:

* Ankle muscle strength (4 directions in concentric and eccentric modes)
* Joint range of motion (ROM)
* Static balance
* Dynamic balance Strength measurements will be assessed using an isokinetic dynamometer (Isomed 2000), joint range of motion using a goniometer, dynamic balance using the Y Balance Test (YBT), and static balance using the Diers Formetric 4D pedobarographic balance system. Strength measurements will be performed at angular velocities of 30°/s and 120°/s for plantar flexion and dorsiflexion and 60°/s and 90°/s for inversion and eversion in both the dancer and control groups.

The primary objective of the study is to determine the relationship between a history of ankle injury and these intrinsic parameters. It also aims to compare the control group with ballet dancers who have not suffered an ankle injury in the last year in terms of these intrinsic parameters.

ELIGIBILITY:
Inclusion Criteria:

* For the Dancer Group:

  1. Be 18 years of age or older
  2. Be a professional or academic-level dancer who has been practicing classical ballet regularly (at least 3 days a week) for the past 3 years
  3. Reside in the province of Izmir
  4. Agree to participate voluntarily and have signed an informed consent form
* For the Control Group:

  1. Be 18 years of age or older
  2. Have no prior dance experience
  3. Not have participated in sports that place specific stress on the ankle area (such as ballet, artistic gymnastics, martial arts, soccer, etc.), even if engaging in regular physical activity
  4. Reside in the province of İzmir
  5. Agree to participate voluntarily and have signed an informed consent form

Exclusion Criteria:

1. Having undergone surgery on the lower extremities within the last 6 months
2. Having a history of diagnosed chronic disease related to the nervous system, vestibular system, or musculoskeletal system (e.g., peripheral neuropathy, MS, rheumatoid arthritis, etc.)
3. Having a physical disability that prevents completion of isokinetic or balance tests
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ballet dancers will be ballet dancers aged 18 and over who live in Izmir and have been dancing professionally for at least 3 years. The control group will consist of participants aged 18 and over who are healthy and have no ankle injuries. Participants will be invited to participate in the study on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Ankle muscle strength | baseline(single assessment session; Day 1)
  Isokinetic peak torque of the ankle muscles will be assessed using an isokinetic dynamometer (Isomed 2000).
  Plantar flexion / dorsiflexion (PF/DF): measured at 30°/s and 120°/s angular velocities, in both concentric and eccentric modes.
  Inversion / eversion (INV/EV): measured at 60°/s and 90°/s angular velocities, in both concentric and eccentric modes.
  Units: Newton-meters (Nm).
Dynamic Balance Ability | baseline(single assessment session; Day 1)
  Dynamic balance: Y-Balance Test (Lower Quarter). Reach distances in the anterior, posteromedial, and posterolateral directions will be normalized to leg length. A composite score will be calculated.
  Units: Reach distances (ANT, PM, PL): centimeters (cm)
  Composite score: percent of leg length (%)
  Directional asymmetries: centimeters (cm)
Range of Motion (ROM) of the Ankle and First Metatarsophalangeal (1st MTP) Joint | Baseline (single assessment session; Day 1)
  Active joint range of motion will be measured with a universal goniometer.
  Ankle: dorsiflexion, plantar flexion, inversion, eversion.
  1st MTP joint: dorsiflexion, flexion
  Units: Degrees (°).
Static Balance Ability | baseline(single assessment session; Day 1)
  Static balance: Center of pressure (CoP) trace length, sway area, and mean CoP velocity will be recorded during 30-second quiet stance (feet hip-width apart) using a pedobarography system.
  Units: Millimeters (mm), square millimeters (mm²), millimeters per second (mm/s).

SECONDARY OUTCOMES:
Strength Ratios | Baseline (single assessment session; Day 1)
  Plantar flexion / dorsiflexion (PF/DF) strength ratio.
  Inversion / eversion (INV/EV) strength ratio. Calculated as the ratio of peak torques obtained from isokinetic testing. Units: Unitless ratio.
Side-to-Side Strength Asymmetry | Baseline (single assessment session; Day 1)
  Calculated for PF/DF and INV/EV. Units: Percentage (%).
Y-Balance Test Asymmetry | Baseline (single assessment session; Day 1)
  Absolute right-left differences in anterior, posteromedial, and posterolateral reach distances.
  Units: Centimeters (cm).

OTHER OUTCOMES:
True Limb Length | Baseline (single assessment session; Day 1)
  Anatomical limb length measured from anterior superior iliac spine to medial malleolus bilaterally.
  Units: Centimeters (cm).
Body Mass Index (BMI) | Baseline (single assessment session; Day 1)
  Height measurements will be converted from centimeters to meters for the calculation. BMI will be calculated as weight (in kilograms) / height (in meters) x height (in meters).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet E ENGİN, Resident, Principal Investigator — Ege University Faculty of Medicine, Department of Sports Medicine; Seçkin Şenışık, assistant professor, Study Chair — Ege University Faculty of Medicine, Department of Sports Medicine
Locations (1):
- Ege University Faculty of Medicine, Department of Sports Medicine,, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plisky PJ, Rauh MJ, Kaminski TW, Underwood FB. Star Excursion Balance Test as a predictor of lower extremity injury in high school basketball players. J Orthop Sports Phys Ther. 2006 Dec;36(12):911-9. doi: 10.2519/jospt.2006.2244. PMID 17193868
- [Background] Zurawski A, Sliwinski Z, Koziel D, Kiebzak W. Monitoring Expression of Balance during Therapy in Children with Postural Disorders. Children (Basel). 2023 May 30;10(6):974. doi: 10.3390/children10060974. PMID 37371206
- [Background] Martin RL, McPoil TG. Reliability of ankle goniometric measurements: a literature review. J Am Podiatr Med Assoc. 2005 Nov-Dec;95(6):564-72. doi: 10.7547/0950564. PMID 16291848
- [Background] Arnold BL, De La Motte S, Linens S, Ross SE. Ankle instability is associated with balance impairments: a meta-analysis. Med Sci Sports Exerc. 2009 May;41(5):1048-62. doi: 10.1249/MSS.0b013e318192d044. PMID 19346982
- [Background] Fong DT, Ha SC, Mok KM, Chan CW, Chan KM. Kinematics analysis of ankle inversion ligamentous sprain injuries in sports: five cases from televised tennis competitions. Am J Sports Med. 2012 Nov;40(11):2627-32. doi: 10.1177/0363546512458259. Epub 2012 Sep 11. PMID 22967824
- [Background] Ramkumar PN, Farber J, Arnouk J, Varner KE, Mcculloch PC. Injuries in a Professional Ballet Dance Company: A 10-year Retrospective Study. J Dance Med Sci. 2016 Mar;20(1):30-7. doi: 10.12678/1089-313X.20.1.30. PMID 27025450
- [Background] Gonosova Z, Linduska P, Bizovska L, Svoboda Z. Reliability of Ankle(-)Foot Complex Isokinetic Strength Assessment Using the Isomed 2000 Dynamometer. Medicina (Kaunas). 2018 Jun 4;54(3):43. doi: 10.3390/medicina54030043. PMID 30344274
- [Background] Nagy P, Brogden C, Greig M. Isokinetic ankle eversion and inversion strength profiling of female ballet dancers. J Sports Sci. 2021 Jan;39(1):1-9. doi: 10.1080/02640414.2020.1803185. Epub 2020 Aug 26. PMID 32844718
- [Background] Lin CW, You YL, Chen YA, Wu TC, Lin CF. Effect of Integrated Training on Balance and Ankle Reposition Sense in Ballet Dancers. Int J Environ Res Public Health. 2021 Dec 3;18(23):12751. doi: 10.3390/ijerph182312751. PMID 34886476
- [Background] Pavlovic M, Ogrinc N, Sarabon N. Body asymmetries as risk factors for musculoskeletal injuries in dancesport, hip-hop and ballet dancers? Eur J Transl Myol. 2022 Nov 28;32(4):11020. doi: 10.4081/ejtm.2022.11020. PMID 36445245
- [Background] Werber B. Dance medicine of the foot and ankle: a review. Clin Podiatr Med Surg. 2011 Jan;28(1):137-54. doi: 10.1016/j.cpm.2010.10.005. PMID 21276523
- [Background] Bowling A. Injuries to dancers: prevalence, treatment, and perceptions of causes. BMJ. 1989 Mar 18;298(6675):731-4. doi: 10.1136/bmj.298.6675.731. PMID 2496824
- [Background] Teitz, C. C. (2000). Hip and knee injuries in dancers. Journal of Dance Medicine & Science, 4, 23-29.
- [Background] Furia JP, Juliano PJ, Wade AM, Schaden W, Mittermayr R. Shock wave therapy compared with intramedullary screw fixation for nonunion of proximal fifth metatarsal metaphyseal-diaphyseal fractures. J Bone Joint Surg Am. 2010 Apr;92(4):846-54. doi: 10.2106/JBJS.I.00653. PMID 20360507
- [Background] Volkova VG, Raisanen A, Benson LC, Ferber R, Kenny SJ. Systematic review of methods used to measure training load in dance. BMJ Open Sport Exerc Med. 2023 Jul 12;9(3):e001484. doi: 10.1136/bmjsem-2022-001484. eCollection 2023. PMID 37457429
- [Background] Smith PJ, Gerrie BJ, Varner KE, McCulloch PC, Lintner DM, Harris JD. Incidence and Prevalence of Musculoskeletal Injury in Ballet: A Systematic Review. Orthop J Sports Med. 2015 Jul 6;3(7):2325967115592621. doi: 10.1177/2325967115592621. eCollection 2015 Jul. PMID 26673541
- [Background] Katakura M, Kedgley AE, Shaw JW, Mattiussi AM, Kelly S, Clark R, Allen N, Calder JDF. Epidemiological Characteristics of Foot and Ankle Injuries in 2 Professional Ballet Companies: A 3-Season Cohort Study of 588 Medical Attention Injuries and 255 Time-Loss Injuries. Orthop J Sports Med. 2023 Feb 28;11(2):23259671221134131. doi: 10.1177/23259671221134131. eCollection 2023 Feb. PMID 36874048
- [Background] Costa MS, Ferreira AS, Orsini M, Silva EB, Felicio LR. Characteristics and prevalence of musculoskeletal injury in professional and non-professional ballet dancers. Braz J Phys Ther. 2016 Jan 19;20(2):166-75. doi: 10.1590/bjpt-rbf.2014.0142. PMID 26786085
- [Background] Wiesler ER, Hunter DM, Martin DF, Curl WW, Hoen H. Ankle flexibility and injury patterns in dancers. Am J Sports Med. 1996 Nov-Dec;24(6):754-7. doi: 10.1177/036354659602400609. PMID 8947396
- [Background] Saleh, H. A. I. A. (2021). Lower limb kinematic analysis to Le Petit Echappé by using two different pointe training pointe and professional pointe in ballet. International Journal of Sports Science and Arts, 17(17), 54-92. https://doi.org/10.21608/eijssa.2020.48542.1054
- [Background] Garrick, J. G. (1999). Early identification of musculoskeletal complaints and injuries among female ballet students. Journal of Dance Medicine & Science, 3(2), 80-83.
- [Background] Bronner S, Ojofeitimi S, Rose D. Injuries in a modern dance company: effect of comprehensive management on injury incidence and time loss. Am J Sports Med. 2003 May-Jun;31(3):365-73. doi: 10.1177/03635465030310030701. PMID 12750128
- [Background] Nilsson C, Leanderson J, Wykman A, Strender LE. The injury panorama in a Swedish professional ballet company. Knee Surg Sports Traumatol Arthrosc. 2001 Jul;9(4):242-6. doi: 10.1007/s001670100195. PMID 11522083
- [Background] Byhring S, Bo K. Musculoskeletal injuries in the Norwegian National Ballet: a prospective cohort study. Scand J Med Sci Sports. 2002 Dec;12(6):365-70. doi: 10.1034/j.1600-0838.2002.01262.x. PMID 12453164
- [Background] Allen N, Nevill A, Brooks J, Koutedakis Y, Wyon M. Ballet injuries: injury incidence and severity over 1 year. J Orthop Sports Phys Ther. 2012 Sep;42(9):781-90. doi: 10.2519/jospt.2012.3893. Epub 2012 Jul 19. PMID 22814244
- [Background] Liederbach M, Dilgen FE, Rose DJ. Incidence of anterior cruciate ligament injuries among elite ballet and modern dancers: a 5-year prospective study. Am J Sports Med. 2008 Sep;36(9):1779-88. doi: 10.1177/0363546508323644. PMID 18753681
- [Background] Shah S, Weiss DS, Burchette RJ. Injuries in professional modern dancers: incidence, risk factors, and management. J Dance Med Sci. 2012 Mar;16(1):17-25. PMID 22390950
- [Background] Russell JA, McEwan IM, Koutedakis Y, Wyon MA. Clinical anatomy and biomechanics of the ankle in dance. J Dance Med Sci. 2008;12(3):75-82. PMID 19618582
- [Background] Russell JA, Shave RM, Kruse DW, Koutedakis Y, Wyon MA. Ankle and foot contributions to extreme plantar- and dorsiflexion in female ballet dancers. Foot Ankle Int. 2011 Feb;32(2):183-8. doi: 10.3113/FAI.2011.0183. PMID 21288419
- [Background] BARNETT CH, NAPIER JR. The axis of rotation at the ankle joint in man; its influence upon the form of the talus and the mobility of the fibula. J Anat. 1952 Jan;86(1):1-9. No abstract available. PMID 14907546
- [Background] Ahonen J. Biomechanics of the foot in dance: a literature review. J Dance Med Sci. 2008;12(3):99-108. PMID 19618585